CLINICAL TRIAL: NCT04271345
Title: Analysis of the Pulmonary Microbiota in a Cohort of Critically Ill Patients Admitted to the Intensive Care Unit. Prospective, Observational Trial.
Brief Title: Lung Microbiota Analysis in Critically Ill Patients Admitted to the Intensive Care Unit.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 1847
Record Dates: First submitted 2019-02-19; First posted 2020-02-17 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Lung Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aims to evaluate the relationship between the heterogeneity of pulmonary microbiota and clinical and outcome variables among critically ill patients admitted to the intensive care unit (ICU). In patients undergoing invasive mechanical ventilation, an aliquot of bronchoalveolar lavage (BAL) fluid will be used in the microbiology laboratory for the analysis of respiratory microbiota through next-generation sequencing technologies and validate computational techniques.

DETAILED DESCRIPTION:
Traditionally, microbiological investigations and clinical trials have contributed to the definition of lower airways as a physiologically sterile district, whose microbiological balance is altered when a respiratory infectious process occur. Actually, the introduction of molecular study methods aiming at the identification of pathogens through genomic sequencing questioned the pardigm of "one bug-one disease", according to which we usually tend to consider a bronchial or pulmonary infectious event as due to the pathogenic role of a single exogenous microorganism. In such a contest, there are truly few data dealing with the characterization of respiratory microbiota in human BAL as well as with the major determinants of this phenomenon and the possible impact on clinical and microbiological outcomes. Our study, although it's a pilot one, aims to evaluate these aspects in a larger cohort of critically ill patients, observing the relationship between the heterogeneity of pulmonary microbiota and clinical and outcome variables. In patients undergoing invasive mechanical ventilation, an aliquot of BAL fluid will be used in the microbiology laboratory for the analysis of respiratory microbiota through next-generation sequencing technologies and validate computational techniques. For each enrolled patient, we will register demographic, clinical and laboratory variables. The benefits deriving from this study lay in the possibility of improving the understanding of characteristics of critical patient's pulmonary microbioma and its clinical impact. Such an information meets the increasingly topical need to customize medical interventions, especially in the context of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* execution of bronchoalveolar lavage sampling, either for clinical indications or in the context of surveillance programs
* acquisition of an informed consent

Exclusion Criteria:

* presence of significant coagulation abnormalities and/or severe respiratory failure
* clearly bloody BAL sample
* small quantity of BAL sample (<5 ml)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICUs and undergoing invasive mechanical ventilation (through oro-tracheal tube or tracheotomy)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Description of the biodiversity of pulmonary microbioma in a cohort of critically ill ICU patients | 36 months
  This aim will be achieved through the use of next-generation sequencing technologies and validate computational techniques, allowing us to taxonomically classify as well as to compare the germs present in BAL samples of ICU patients

SECONDARY OUTCOMES:
Clinical cure, defined by the discontinuation (> 72 hours) from mechanical ventilation | 36 months
  Relate composition and biodiversity of pulmonary microbioma with the occurence and time of clinical cure
Microbiological eradication, defined by a sterile BAL | 36 months
  Relate composition ad biodiversity of pulmonary microbioma with the occurrence and time of microbiological eradication
Duration of mechanical ventilation, in days | 36 months
  Relate composition ad biodiversity of pulmonary microbioma with the duration of mechanical ventilation
Duration of cathecolamins administration, in days | 36 months
  Relate composition ad biodiversity of pulmonary microbioma with the duration of cathecolamins administration
Hospital and ICU lenght of stay, in days | 36 months
  Relate composition ad biodiversity of pulmonary microbioma with hospital and ICU lenght of stay
Mortality at 28 and 90 days | 36 months
  Relate composition ad biodiversity of pulmonary microbioma with mortality at 28 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro De Pascale, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS
Locations (1):
- Fondazione Policlinico A. Gemelli IRCCS, Rome, Italy

REFERENCES:
- [Derived] De Pascale G, Posteraro B, De Maio F, Pafundi PC, Tanzarella ES, Cutuli SL, Lombardi G, Grieco DL, Franchini E, Santarelli G, Infante A, Sanguinetti M, Antonelli M. Lung microbiota composition, respiratory mechanics, and outcomes in COVID-19-related ARDS. Microbiol Spectr. 2024 Apr 2;12(4):e0357423. doi: 10.1128/spectrum.03574-23. Epub 2024 Mar 11. PMID 38466118